CLINICAL TRIAL: NCT00589992
Title: Atrial Fibrillation Mechanism Analysis Through Ibutilide Administration During Pulmonary Vein Ablation.
Brief Title: Ibutilide Administration During Pulmonary Vein Ablation
Acronym: IBAD-AFIB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ball Memorial Hospital (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Antonio Navarrete, MD, Medical Consultants, P.C.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BMH study #762
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Atrial Fibrillation; Pulmonary Vein Ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — ibutilide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ibutilide fumarate — During scheduled radio frequency ablation for atrial fibrillation patients will be infused with 1mg of ibutilide over 10 minutes.

SUMMARY:
To test the hypothesis that localized functional reentry maintains Afib in humans, ibutilide will be administered intravenously in patients undergoing an Afib ablation. The hypothesis of this study is that ibutilide will decrease the high frequency signals observed in Afib suggesting the presence of micro reentrant circuits as the basic mechanism of Afib, especially for the paroxysmal Afib group. The potential difference in response to the ibutilide in patients with paroxysmal versus persistent Afib may show the difference in the underlying mechanism of Afib between these two groups.

ELIGIBILITY:
Inclusion Criteria:

* patients to be scheduled for atrial fibrillation radio frequency ablation
* paroxysmal, permanent symptomatic atrial fibrillation refractory to conventional treatment
* symptomatic atrial fibrillation that do not want or desire to take medication or undergo cardioversion
* patients on antiarrhythmics that can be discontinued 5 half lifes prior to the procedure except for Amiodarone

Exclusion Criteria:

* patients with recent major hemorrhage (within 6 months)
* patients with a coagulopathy
* patients who are pregnant or breast feeding
* patients with acute congestive heart failure
* patients with hypokalemia or hyperkalemia
* patients with a prolonged QTc > 440mms
* patients with polymorphic ventricular tachycardia secondary to antiarrhythmic class III and class I
* patients with left ventricular dysfunction < 40%
* patients with a history of recent MI (< 1 month)
* patients with a history of an angioplasty of < 1 month
* patients with a history of coronary artery bypass grafting surgery of < 3 months.
* patients with a history of chronic renal failure or a creatinine clearance of < 30ml/m
* patients with a history of stroke of < 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-10; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
To discern the basic mechanism of Afib by studying its response to Ibutilide administration. | one year

SECONDARY OUTCOMES:
To compare the ibutilide response in patients with paroxysmal versus permanent Afib | one year
To study the subgroup of patients that converted to sinus rhythm in order to identify various factors that may have increased their susceptibility to ibutilide. | one year
To improve the current results of pulmonary vein isolation by performing a procedure guided by ablation of high dominant frequency areas. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Navarrete, MD, Principal Investigator — Staff Physician, Ball Memorial Hospital
Locations (1):
- Medical Consultants, P.C., Muncie, Indiana, United States